CLINICAL TRIAL: NCT02894619
Title: Assessment of the Prevalence and Severity of Urinary and Ano-rectal Functional Disorders and Their Impact on Quality of Life and Sexuality on CF Adults of the North-West CF Network
Brief Title: Urinary and Anorectal Functional Disorders and Their Impact on CF Adults (PerineoMucoRMO)
Acronym: PerineoMuco
Status: Completed | Type: Observational
Sponsor: Fondation Ildys (Other)
Collaborators: Vaincre la Mucoviscidose (Other); University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ILDYS-ISRNI-2015003; RC20160501608 (Other Grant/Funding Number: Vaincre La Mucoviscidose (CF French Association))
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis
Keywords: urinary incontinence; anal incontinence; sexuality; quality of life
MeSH Terms: conditions — Cystic Fibrosis; Urinary Incontinence; Encopresis; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study evaluates prevalence of functional perinea disorders (stress urinary incontinence, overactive bladder syndrome, dysuria, anal incontinence) on CF adults patients of the North-West CF Network. Its aims are to measure the severity of urinary and anorectal symptoms ; assess their impact on patients' quality of life, sexuality, care and social life and relationships ; identify the medical and demographic factors associated with the severity of urinary and anorectal disorders and their impact and determine the relationship between the severity of these disorders, various repercussions, and risk factors.

DETAILED DESCRIPTION:
Urine and/or anal leakage are more frequent and troublesome for CF patients: leaks occur during efforts or laugh like in other people, but also when coughing or sneezing, which are amplified during periods of exacerbation and with the degradation of the pulmonary condition. In addition, fear of leakage can disrupt medical care: discomfort during physiotherapy, pulmonary function test. Urinary and anorectal functional disorders are therefore not only a factor degrading the quality of life but also a risk factor for worsening bronchial obstruction, patients limiting their cough and / or their care to avoid episodes of leakage. Given the lack literature data, investigators wanted to explore these areas.

Validated and specific questionnaires will be self and anonymously administered to adult patients (n=175). The time requested to fill the forms is estimated to 1H. Questionnaires about sexual health are optional.

Prospects considered, depending on the results, are:

* Extension to the adolescent population (14 and over);
* National extension;
* Systematic proposal of a screening and an appropriate management of pelvic floor functional disorders, depending on influent characteristics (age, gender ...): multidisciplinary working group to develop guidelines and specific tools for professional training and / or patient education;
* Implementation of a comparative study of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and over
* Cystic fibrosis confirmed by sweat test or genetic
* Followed in an adult or mixed CF Center of the French North-West CF Network
* Not transplanted and not entered on the waiting list for transplantation
* In a stable condition for at least 4 weeks
* Able to understand and respect the protocol and its requirements
* Who signed the consent prior to any other procedure protocol

Exclusion Criteria:

* Major patients under guardianship / curatorship
* Patients seen in emergency situation
* Pregnant patients
* Dialysis patients
* Patients with urolithiasis
* Patients with severe exacerbation at the time of inclusion
* Patients on intravenous antibiotics within 4 weeks prior to inclusion
* Patient with an urinary tract infection (evaluation by dipstick at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CF adults patients of the French North-West CF Network
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Urinary Symptom Profile (USP) score | at time of inclusion
  Assesses lower urinary tract symptoms (stress urinary incontinence, overactive bladder syndrome and dysuria)

SECONDARY OUTCOMES:
Wexner Fecal Incontinence Scale | at time of inclusion
  Assesses anal incontinence and its impact on quality of life
SF-Qualiveen questionnaire | at time of inclusion
  Assesses impact of urinary disorders on quality of life
Cystic Fibrosis Questionnaire-Revised (CFQ-R) | at time of inclusion
  Assesses quality of live related to cystic fibrosis
International Index of Erectile Function (IIEF5) questionnaire | at time of inclusion
  Assesses male sexual dysfunction
Female Sexual Function Index (FSFI) | at time of inclusion
  Assesses female sexual dysfunction

OTHER OUTCOMES:
Informations Questionnaire | at time of inclusion
  identification and prevalence of risk factors; impact degree of disorders on care, social and love life, sexuality

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Ramel, MD, Study Director — Fondation Ildys; Katelyne Hubeaux, MD, Study Director — Fondation Ildys
Locations (6):
- France (6):
  - CF Center - University Hospital, Angers
  - CF Center - Hôpital Laennec, Nantes
  - CF Center - Hopital Pontchaillou, Rennes
  - CF Center - Fondation Ildys Site de Perharidy, Roscoff
  - CF Center - Groupe Hospitalier Sud Réunion, Saint-Pierre-des-Corps
  - CF Center - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Informations aboit project — http://www.reseau-muco-ouest.fr/projets/22-perineomuco